CLINICAL TRIAL: NCT00677547
Title: Humoral and Cell-mediated Immune Response to Influenza Vaccine in Kidney Tranpslant Recipients.
Brief Title: Cell-mediated Immune Response to Influenza Vaccine
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Assistant Professor of Medicine, University of Alberta
Other Study IDs: 7061
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Kidney Transplant
Keywords: Kidney; Influenza vaccine; CMI
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Kidney transplant recipients
- 2: Healthy volunteers

SUMMARY:
Influenza virus is an important cause of morbidity in the transplant population and can lead to viral and bacterial pneumonia. Although the annual influenza vaccine is recommended for organ transplant patients, studies have shown that the standard inactivated influenza vaccine has poor immunogenicity in this population. One major hurdle in the evaluation of the response of influenza vaccine in immunocompromised patients is the lack of correlation between humoral response and efficacy of the vaccine. In patients with poor immune responses, cellular immunity may have a better correlation than humoral immunity with vaccine protection. We plan to assess the utility of 3 assays that evaluate the cell-mediated immune response (granzyme B, interleukin-10 (IL-10), and interferon-gamma (IFN-)) after influenza vaccine in kidney transplant recipients. Results from this study have the potential to directly improve patient care. The new monitoring assays may more accurately determine the risk for development of influenza infection, and therefore allowing a better prevention strategy.

DETAILED DESCRIPTION:
There is limited prospective data on influenza infections in transplant recipients. However, influenza can be a significant cause of morbidity and mortality in some organ transplant populations. Reported attack rates have varied considerably and are likely due to differences in transplant populations, immunosuppression protocols, exposures, and type and virulence of circulating influenza viruses. Complications of influenza infection appear to be common in solid organ transplant (SOT) populations. There appears to be a relatively high rate of progression to viral pneumonia in some reports especially in lung transplant recipients. In one study of organ transplant recipients over a 10-year period, the rate of influenza infection ranged from 2.8 cases/1000 person years (liver transplant) to 41.8 cases/1000 person years (lung transplant). Complications including secondary bacterial pneumonia (17%) as well as extrapulmonary complications such as myocarditis, and myositis were observed. Influenza (and other respiratory viral infections) may lead to important immunological sequelae resulting in graft rejection and/or graft dysfunction. This may be secondary to activation of immunological mechanisms, including the upregulation of pro-inflammatory cytokines such as TNF-α, IL-6 and IL-8. Some studies of kidney and liver recipients have reported a high incidence of acute rejection following infection with influenza. However, while associations between influenza infection and rejection have been reported, a causal relationship has yet to be established.

Influenza vaccination has become the standard of care for several population groups. The Centers for Disease Control and Prevention (CDC) and the Canadian National Advisory Committee on Immunization (NACI) currently recommends this vaccine for children > 6 months, healthy adults, the elderly and all immunocompromised patients such as those with organ transplants (www.cdc.gov). The currently available influenza vaccine is a subunit vaccine containing the purified surface glycoproteins of the virus, hemagglutinin and neuraminidase. The vaccine contains 15g antigen from each of 2 circulating subtypes of influenza A and 15 g of an influenza B subtype (www.who.int). The vaccine is administered by the intramuscular route, generally in the deltoid muscle in adults. The standard dose is 0.5 mL.

Annual influenza vaccination is currently considered the main strategy to prevent influenza infection for all organ transplant recipients. However, a large number of studies have shown that the immunogenic response to this vaccine is suboptimal and ranges from 15-70%. This number varies depending on the organ transplanted and the immunosuppressive regimen used. Indeed, some studies in kidney transplant recipients, especially in the pediatric population, have shown similar responses to the influenza vaccine than in healthy controls.

Monitoring of immune response to influenza vaccine. Laboratory monitoring of response to influenza vaccine can be done by hemagglutination inhibition assay. Although laboratory serology is a surrogate marker for protection, it is widely used. This is primarily due to the large numbers of patients that would be needed to show vaccine efficacy if documented influenza infection were used as the outcome. The HIA is also used by the World Health Organization to validate annual vaccines. However, it is not known if the criteria used for the general population may be applied in immunocompromised patients. In fact, in the elderly it has been clearly proved that the standard cutoff for antibody levels of 40 units did not protect against influenza. In a study with 397 elderly vaccinated against influenza, 60% of persons who developed influenza had an antibody level of 40 units. To our knowledge, the absolute titer of antibody required to confer significant protection from illness is unknown in transplant patients.

Cell-mediated immunity after influenza vaccination. Recently, specific cellular responses have also been implicated in protection against influenza, independently of the humoral response. Cellular mediated immunity has been evaluated measuring IL-2 and IFN-(for T-helper type 1 response), IL-10 (for T-helper type 2 response), and granzyme B expression (which correlates with lytic activation). The cell-mediated immune response has been mainly used to evaluate the response to influenza vaccine in the elderly. In a study with 90 persons >60 year-old, the IFN-/IL-10 ratio and granzyme B levels were significantly higher in persons who did not develop influenza during the follow-up, compared to persons who developed influenza. There was no correlation between the antibody levels and the risk of developing influenza infection. In a previous study, granzyme B levels were found to be higher in young people than in old people. Taken together, these data suggest that cell-mediated immune response may correlate better with the risk of influenza after vaccination.

The cell-mediated immune response after influenza vaccine has been only assessed in one study involving solid organ recipients. Mazzone et al. evaluated in 43 lung transplant recipients and in 21 healthy controls. IL-2, IL-10, IFN-, and granzyme B levels did not increase from pre- to post-vaccination in the lung transplant group. Both pre- and post-cytokine levels were lower in the transplant group compared to the control group.

The study we propose is a prospective cohort trial designed to assess the immunogenicity after a standard influenza vaccination measuring the cellular immunity in a cohort of kidney transplant recipients, and correlate it with the standard humoral immunity.

ELIGIBILITY:
Adult kidney transplant recipients:

Inclusion Criteria:

* Age ≥ 18
* Greater than 3 months post-transplant

Exclusion Criteria:

* Egg allergy
* Previous life-threatening reaction to influenza vaccine (ie Guillain Barre Syndrome)
* On anticoagulants such as warfarin that precludes intramuscular injection
* Ongoing therapy for rejection
* Febrile illness in the past two weeks
* Unable to provide informed consent

Healthy volunteers

Inclusion Criteria:

- Age ≥ 18

Exclusion Criteria:

* Egg allergy
* Previous life-threatening reaction to influenza vaccine (ie Guillain Barre Syndrome)
* On anticoagulants such as warfarin that precludes intramuscular injection
* On immunosuppressive medication (prednisone, immunomodulators for autoimmune diseases)
* Underlying autoimmune disease (eg, sarcoid, lupus, rheumatoid arthritis, Crohn's disease)
* Febrile illness in the past two weeks
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients and healthy volunteers (enrolled among hospital staff)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Correlation between the levels of Granzyme B and the IFN-/IL-10 ratio and the humoral response (HIA titers of 1:40, or serological response with a four-fold or greater increase in HI antibody titers), in the transplant and the control groups. | 3 months

SECONDARY OUTCOMES:
Local and systemic adverse events to vaccination. Rates of allograft rejection in the 6 months following vaccination Documented influenza infection (by direct fluorescent antibody, viral culture, or PCR) in the 6 months following vaccination | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Ison MG, Hayden FG. Viral infections in immunocompromised patients: what's new with respiratory viruses? Curr Opin Infect Dis. 2002 Aug;15(4):355-67. doi: 10.1097/00001432-200208000-00002. PMID 12130931
- [Background] Ljungman P, Andersson J, Aschan J, Barkholt L, Ehrnst A, Johansson M, Weiland O. Influenza A in immunocompromised patients. Clin Infect Dis. 1993 Aug;17(2):244-7. doi: 10.1093/clinids/17.2.244. PMID 8399875
- [Background] Kumar D, Erdman D, Keshavjee S, Peret T, Tellier R, Hadjiliadis D, Johnson G, Ayers M, Siegal D, Humar A. Clinical impact of community-acquired respiratory viruses on bronchiolitis obliterans after lung transplant. Am J Transplant. 2005 Aug;5(8):2031-6. doi: 10.1111/j.1600-6143.2005.00971.x. PMID 15996256